CLINICAL TRIAL: NCT07373353
Title: AMJ-401 Japan Clinical Trial
Brief Title: A Clinical Evaluation of AMJ-401
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10615
Record Dates: First submitted 2026-01-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Heart Disease (IHD)
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/Treatment (Experimental)
  Interventions: Device: AMJ-401

INTERVENTIONS:
Device: AMJ-401 — Patients undergoing percutaneous coronary intervention of one or two de novo native coronary artery lesions with AMJ-401 in separate epicardial coronary vessels

SUMMARY:
A Clinical Evaluation of AMJ-401 in the Treatment of Subjects with Ischemic Heart Disease in Japan

DETAILED DESCRIPTION:
The objective of this clinical investigation is to demonstrate the safety and performance of AMJ-401 Everolimus Eluting Resorbable Scaffold System in the treatment of de novo native coronary artery lesions. Patients undergoing percutaneous coronary intervention of one or two de novo native coronary artery lesions in separate epicardial coronary vessels will be evaluated.

ELIGIBILITY:
Inclusion Criteria

1. Subject must be at least 18 years of age.
2. Subject or a legally authorized representative must be able to provide written Informed Consent prior to any study related procedure, per site requirements.
3. Subject must have evidence of myocardial ischemia (e.g., stable angina, silent ischemia, unstable angina, acute myocardial infarction) suitable for elective PCI.
4. Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Subject must be able to take dual antiplatelet therapy (DAPT) for minimum of 12 months following the index procedure and anticoagulants prior/during the index procedure, and the subject has no known allergic reaction, hypersensitivity or contraindication to aspirin, clopidogrel, prasugrel, ticagrelor, ticlopidine or heparin.
6. Female subjects of childbearing potential must not be pregnant* at screening and do not plan pregnancy for at least 12 months following the index procedure.

   * Female subjects of child-bearing potential must have a negative pregnancy result within 7 days prior to the index procedure.
7. Female subjects must not be breast-feeding at the time of the screening visit and will not be breast-feeding for at least 12 months following the index procedure.
8. Subject agrees to not participate in any other investigational or invasive clinical study for a period of 13 months following the index procedure.

Exclusion Criteria:

1. Elective surgery planned within 12 months after the procedure that will require general anesthesia or discontinuing either aspirin or P2Y12 inhibitor.
2. Subject has known hypersensitivity or contraindication to device material and its degradants (everolimus, PLLA, PDLLA, platinum, lactic acid, and lactide) that cannot be adequately pre-medicated.
3. Subject has a known contrast sensitivity that cannot be adequately pre-medicated.
4. Subject with known diagnosis of ST-elevation myocardial infarction (STEMI) within 72 hours of the index procedure.
5. The subject is currently experiencing clinical symptoms consistent with new onset acute myocardial infarction (AMI), such as nitrate-unresponsive prolonged chest pain with ischemic ECG changes.
6. Subject has an unstable cardiac arrhythmia which is likely to become hemodynamically unstable due to their arrhythmia
7. Subject has a known left ventricular ejection fraction (LVEF) < 30% (LVEF may be obtained at the time of the index procedure prior to subject registration if the value is unknown and the site Investigator believes it is necessary).
8. The target vessel was treated by PCI within 12 months prior to index procedure.
9. Prior PCI within the non-target vessel is acceptable if performed anytime > 30 days before the index procedure, or between 24 hours and 30 days before the index procedure if successful and uncomplicated.
10. Subject requires future staged PCI either in target or non-target vessels.
11. Subject has a malignancy that is not in remission.
12. Subject is receiving immunosuppressant therapy or has known life-threatening immunosuppressive or life-threatening autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.). Note: corticosteroids are not included as immunosuppressant therapy, diabetes mellitus is not regarded as autoimmune disease.
13. Subject has received any solid organ transplants or is on a waiting list for any solid organ transplants.
14. Subject has previously received or scheduled to receive radiotherapy to coronary artery (brachytherapy), or chest/mediastinum.
15. Subject is receiving or will require chronic anticoagulation therapy (e.g., warfarin).
16. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3.
17. Subject has documented or suspected cirrhosis of Child-Pugh ≥ Class B.
18. Subject has known renal insufficiency:

    * Dialysis at the time of screening or
    * An estimated GFR < 30 ml/min/1.73m2
19. Subject has a high risk of bleeding, or;

    * Subject has a history of bleeding diathesis or coagulopathy.
    * Subject has had a significant gastro-intestinal or significant urinary bleed within the past six months.
    * Subject has prior intracranial bleed (including severe permanent neurologic deficit that seems to be caused by previous intracranial bleeding).
    * Subject has known intracranial pathology that may cause intracranial bleeding per investigator assessment (e.g., untreated aneurysm greater than 5 mm, arteriovenous malformation)
    * Subject will refuse blood transfusions.
    * Subject is receiving antiplatelet medication other than aspirin or P2Y12 inhibitor for the treatment of another condition and cannot discontinue them
20. Subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past six months,
21. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion via any vessel.
22. Subject has life expectancy < 3 years.
23. Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason.
24. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
25. Subject whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., subordinate hospital staff or sponsor staff).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Acute Strut Fracture | 6 months
  Acute strut fracture is assessed on a per-subject basis per final post-procedure OCT.
Strut Coverage | 6 months
  Strut coverage is assessed at 6-month OCT follow-up exam as the rate of uncovered struts on a per strut basis.

CONTACTS AND LOCATIONS:
Locations (1):
- Mitsui Memorial Hospital, Tokyo, Chiyoda-ku, Japan

IPD SHARING:
Plan to Share IPD: Undecided